CLINICAL TRIAL: NCT02505451
Title: Comprehensive Analysis of Regional Myocardial Function in Response to Dobutamine Stress in Metabolic Syndrome and Type 2 Diabetic Patients. Effect of Cardiac Adiposity, Inflammation and Hyperglycaemia
Brief Title: Myocardial Regional Function by Dobutamine Stress Echocardiography in the Metabolic Syndrome and Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Avignon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UAPV-022015-SFC
Record Dates: First submitted 2015-07-03; First posted 2015-07-22 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Diabetes-related Complications
Keywords: Metabolic syndrome; diabetes; myocardial function; dobutamine
MeSH Terms: conditions — Diabetes Complications; Metabolic Syndrome; Diabetes Mellitus | interventions — Dobutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Type 2 diabetic patients (Experimental): Regional myocardial function will be assessed during dobutamine stress echocardiography in asymptomatic patients with type II diabetes (according to the American Diabetes Association, 2012) free of coronary diseases.
  Interventions: Drug: dobutamine
- Metabolic syndrom (Experimental): Regional myocardial function will be assessed during dobutamine stress echocardiography in asymptomatic patients with the Metabolic syndrome (according to Alberti et al 2009) free of diabetes and coronary diseases.
  Interventions: Drug: dobutamine
- controls (Experimental): Regional myocardial function will be assessed during dobutamine stress echocardiography in healthy subjects.
  Interventions: Drug: dobutamine

INTERVENTIONS:
Drug: dobutamine — In each participant, dobutamine will be administered via intravenous infusion in doses of 10, 20, 30 and 40 lg/kg/min during 3-min stages and 2D strain echocardiography will be performed at each stage.

SUMMARY:
Summary.

Theoretical Rationale:

The left ventricular myocardial performance results from a complex interplay between linear deformations (longitudinal, circumferential and radial) and twist/ untwist mechanics. These components of myocardial mechanics can be assessed, at rest and during stress conditions, by high resolution echocardiography using the "2D-strain" technology and constitute good indexes of tissue intrinsic contractility / relaxation properties. Type 2 diabetes (T2DM) and metabolic syndrome (MS) are associated with an increased risk for cardiac diseases. While several clinical studies have reported, particularly in T2DM, a diastolic dysfunction (concept of "diabetic cardiomyopathy"), the existence of impaired regional myocardial function, with altered intrinsic contractility properties, remains largely unanswered, especially in the SM. Stress echocardiography is very interesting to reveal myocardial dysfunction, discrete or absent at rest. To the best of our knowledge, no scientific study is, however, today available on the kinetics of linear strains and twist/untwist dynamics in response to stress in T2DM as well as SM. The epicardial adipose tissue is the source of production of important pro-inflammatory cytokines that have the potential, through an exacerbation of oxidative stress, to impair coronary endothelial function, increase fibrosis, but also directly affect cardiomyocyte calcium homeostasis. An increase in epicardial adipose tissue is consensually reported in T2DM and SM and is clearly associated with coronary atherosclerosis. A link between cardiac adiposity and overall cardiac function, particularly diastolic, is now suggested but to our knowledge no study has challenged its association with myocardial dysfunction in T2DM as SM patients.

Objectives and Methodology: - To investigate regional myocardial linear deformations and torsion, at rest and in response to a dobutamine stress, in asymptomatic T2DM and SM patients without clinical complications, - to study the links between expected regional myocardial abnormalities and inflammation, hyperglycemia and cardiac adiposity. A control group of healthy individuals matched for sex and age will also be included.

All the subjects will benefit from a clinical, anthropometric and biological evaluation. In addition, conventional echocardiography (remodelling and global diastolic and systolic functions) complemented by a functional analysis by tissue Doppler imaging will be performed. Furthermore, 2D cine loops will be recorded in the apical 4, 3 and 2- chamber views for the objective assessment of myocardial longitudinal deformations as well as in the parasternal short axis (base and apex) for the evaluation of the circumferential deformations and basal and apical rotations and left ventricular torsion, at rest and under low dose of dobutamine (110 and 120 bpm).

ELIGIBILITY:
Inclusion Criteria:

* Male and female 40-65 years old, asymptomatic and free of coronary disease

Exclusion Criteria:

* for all the subjects :
* body mass index > 35 kg / m2, defining severe obesity,
* Under insulin therapy,
* Poorly controlled hypertension (> 140/95)
* Peripheral vascular disease (> stage II of Leriche)
* Heart disease or known coronary artery disease,
* Known and poorly compensated thyroid dysfunction,
* Nocturnal apnea syndrome,
* Inability to give written informed consent,
* Chronic diseases,
* moderate to severe left ventricular hypertrophy :> 109 g / m2 in women and> 132 g / m2 in men and parietal thickness > 13mm.

for the diabetic patients only :

* poor glycemic control (HbA1c > 9%)
* severe autonomic or peripheral neuropathy,
* Severe diabetic retinopathy,
* Advanced Diabetic nephropathy (defined by documented proteinuria and / or renal failure).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Regional longitudinal strain | day 1
  Regional myocardial function will be evaluated for each participant at rest and during low dose dobutamine within a single session.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Obert, PhD, Study Director — Laboratory of Cardiovascular Pharm-Ecology, Faculty of Health and Sciences, university of Avignon, 33 rue louis pasteur 84000 Avignon, France.
Locations (1):
- Hospital Henri Duffaut, Avignon, PACA, France